CLINICAL TRIAL: NCT04943393
Title: Remote Assessment of Working Memory and Anxiety in Individuals With Early-Treated Phenylketonuria (PKU)
Brief Title: Remote Neurocognitive and Psychological Assessment in PKU
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Shawn Christ, Associate Professor, University of Missouri-Columbia
Other Study IDs: 2034504
Record Dates: First submitted 2021-06-02; First posted 2021-06-29 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood phe levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with PKU: Adults with early-treated PKU
  Interventions: Other: nointervention
- Individuals without PKU: Adults without PKU who are otherwise healthy
  Interventions: Other: nointervention

INTERVENTIONS:
Other: nointervention — Nointervention

SUMMARY:
PKU is a rare autosomal recessive condition associated with disruption in dopamine synthesis. Although early diagnosis and treatment prevent the severe impairments associated with untreated PKU, individuals with early-treated PKU (ETPKU) nonetheless experience significant sequelae, including impaired working memory and increased risk for anxiety problems. Past research with other clinical populations (e.g., generalized anxiety disorder) suggests that the two phenomena may be linked, with increased anxiety contributing to poorer WM performance. Currently we propose to initiate an exciting new line of research examining the potential relationship between anxiety and WM in ETPKU. The proposed study will also apply remote neuropsychological performance-based assessment to the study of ETPKU and thus overcoming the geographical limitations/challenges associated with recruitment of participants with this rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants with PKU will be included if they were diagnosed as newborns and immediately started on treatment.

Exclusion Criteria:

* Individuals with a history of neurologic compromise or major medical disorder unrelated to PKU (e.g., closed head injury, diabetes, multiple sclerosis) will be excluded. In addition, individuals with PKU will be excluded if they are on a medication called Peg-Valiant/ PEG-PAL/ Pegvaliase/Palynziq.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals age 18-40 years old with and without PKU
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Working Memory performance | 2.5-3 hrs total over approx 1-3 weeks
  Composite score based on multiple working memory-related CANTAB tests

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Christ, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: Undecided
To be determined